CLINICAL TRIAL: NCT00449787
Title: A Randomized Clinical Trial to Compare Naproxen and Sumatriptan for Headache Patients Discharged From the Emergency Department (ED)
Brief Title: Comparing Naproxen to Sumatriptan for Emergency Headache Patients
Acronym: HEDNet2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin W. Friedman, MD, Associate professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-11-472
Record Dates: First submitted 2007-03-19; First posted 2007-03-21 (Estimated); Results first posted 2012-11-29 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Migraine; Tension-type Headache; Primary Headache Disorder
Keywords: Emergency department; headache; migraine
MeSH Terms: conditions — Migraine Disorders; Tension-Type Headache; Headache Disorders, Primary; Emergencies; Headache | interventions — Sumatriptan; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sumatriptan (Active Comparator): Sumatriptan 100 mg tablet
  Interventions: Drug: Sumatriptan 100 mg
- Naproxen (Active Comparator): Naproxen 500 mg tablet
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: Sumatriptan 100 mg — Sumatriptan 100mg tablet
  Arms: Sumatriptan
Drug: Naproxen — Naproxen 500mg tablet
  Arms: Naproxen

SUMMARY:
2/3 of patients discharged from an emergency department after treatment for an acute headache will still be bothered by headache within 24 hours of emergency department (ED) treatment. The goal of this study is to compare two medications, naproxen and sumatriptan, to determine which is better for the treatment of recurrent headache within 24 hours of emergency department discharge.

DETAILED DESCRIPTION:
Two-thirds of the five million headache patients who present to US emergency departments (ED) annually are suffering an acute exacerbation of a primary headache disorder. Of these acute primary headaches, migraine is the most frequently encountered disease entity in the ED, accounting for 60% of primary headaches, followed by tension-type headaches, which represent 10% of all primary headaches seen in the ED. About ¼ of all acute primary headaches seen in the ED cannot readily be given a specific diagnosis3. Multiple parenteral treatments are used to treat acute primary headaches1, but to date, regardless of specific headache diagnosis, no medication eliminates the frequent recurrence of headache after ED discharge. To date, it is unknown which medication patients should be given when discharged from an ED after treatment for a primary headache. This study will compare two oral headache treatments to determine which one relives pain more effectively.

Specific aims:

1) To determine which of two oral medications is more efficacious for all acute primary headache patients who are discharged from an ED.

Primary hypotheses:

In the 48 hour period following ED treatment for a primary headache, sumatriptan 100mg will relieve pain better than naproxen 500mg, as measured by an 11-point numerical rating scale for pain.

ELIGIBILITY:
Inclusion Criteria:

* Treated in the emergency department for acute primary headache

Exclusion Criteria:

* Allergy, intolerance, or contra-indication to one of the study medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2007-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W. Friedman, MD,MS, Principal Investigator — Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York

REFERENCES:
- See also: Study manuscript posted on Pubmed Central — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2902611/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sumatriptan | Naproxen
Started | 203 | 198
Completed | 98 | 98
Not Completed | 105 | 100
Not completed — Lost to Follow-up | 10 | 8
Not completed — Did not require medication | 95 | 92

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sumatriptan | Naproxen | Total
Number analyzed (Participants) | 203 | 198 | 401
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (10) | 35 (10) | 36 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 168 | 341
  Male | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Scale
Description: Within 48 hours of ED discharge, participants were allowed to take the investigational medication. At the moment they took the investigational medication, they were asked to record a number from 0 to 10, which represented their headache. 0 signified no pain and 10 signified the worse pain imaginable.
  Two hours later, participants were asked again to record their pain on a scale from 0 to 10. The outcome is the change in pain between baseline and two hours and will be a number between 0 and 10. Greater numbes signify greater relief
Time Frame: Baseline, two hours
Population: After discharge from the emergency room, some patients had headache requiring use of medication and some did not. Only those patients who took the investigational medication were included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sumatriptan: Sumatriptan 100mg tablet
Arm/Group | Sumatriptan | Naproxen
Number analyzed (Participants) | 98 | 98
units on a scale | 4.1 (3.1) | 4.3 (3.0)

2. Secondary Outcome: Headache-related Functional Disability
Description: This is a recommend outcome in headache research. At the time of the assessment (48 hours after ER discharge), patients are asked to report their current level of functional impairment: severe (unable to do any activities); moderate (able to do a few activities); mild (able to do many but not all activities) or none (able to do all activities). For this analysis, patient's answers were dichotomized into some impairment or no impairment.
Time Frame: Baseline, two hours
Population: Patients who reported any level of functional impairment (mild, moderate, or severe) are tabulated here.
Measure: Number; unit: participants
Arm/Group | Sumatriptan | Naproxen
Number analyzed (Participants) | 98 | 97
participants | 41 | 36

3. Secondary Outcome: Patient Satisfaction
Description: At the 48 hour assessment, patients were asked, "The next time you go to an emergency room with a headache, do you want to receive the same medication". This outcome tabulates the number of affirmative responses.
Time Frame: 48 hours after ER discharge
Measure: Number; unit: participants
Arm/Group | Sumatriptan | Naproxen
Number analyzed (Participants) | 92 | 96
participants | 69 | 68

ADVERSE EVENTS:
Arm/Group | Sumatriptan | Naproxen
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/98
Other Adverse Events (participants affected / at risk) | 25/97 | 18/97
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sumatriptan (N=97) | Naproxen (N=97)
Other (Musculoskeletal and connective tissue disorders) | 12 (12) | 0 (0) — Various non-serious adverse events including myalgia, facial pains, and non-specific complaints
Gastrointestinal complaint (Gastrointestinal disorders) | 9 (9) | 7 (7) — nausea, vomiting, epigastric pain, or diarrhea
Neurological (Nervous system disorders) | 4 (4) | 11 (11) — Dizzy, lightheaded, non-specific weakness, drowsy, headache

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No